CLINICAL TRIAL: NCT07094321
Title: Predicting Postoperative Myocardial Injury: A Retrospective Cohort Study Comparing Absolute Versus Relative Definitions of Intraoperative Hypotension
Brief Title: Study on the Correlation Between Intraoperative Hypotension and Postoperative Myocardial Injury
Status: Active, not recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Kan Wang, Dr, China-Japan Friendship Hospital
Other Study IDs: ChinaJapanFH
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Injury After Noncardiac Surgery (MINS); Hypotension During Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MINS group: Patients who experienced postoperative cardiac dysfunction
- Non-MINS group: Patients who did not experience postoperative cardiac dysfunction

SUMMARY:
The investigators are conducting an important study aimed at better understanding and predicting a potential complication after non-cardiac surgery: myocardial injury. This research is crucial for enhancing surgical safety and improving patient outcomes.

Simply put, postoperative myocardial injury (PMI) means that heart muscle cells are damaged after non-cardiac surgery. While it might not cause obvious chest pain like a heart attack, it can show up as abnormalities on an electrocardiogram (ECG) or in blood tests (like elevated troponin levels). This type of injury is a significant factor contributing to postoperative complications and even mortality.

During surgery, hypotension-or low blood pressure-is a common occurrence. The investigators know that maintaining adequate blood pressure is essential for the heart to receive a sufficient blood supply. If blood pressure drops too low, the heart's blood supply can be reduced, potentially leading to oxygen deprivation and damage to heart muscle cells.

While it's widely accepted that low blood pressure is linked to myocardial injury, precisely defining "low blood pressure" during surgery has been a persistent challenge.

* Historically, the investigators have focused on the "absolute value" of blood pressure, such as a fixed mean arterial pressure (MAP) threshold (e.g., below 65 mmHg). Many studies have indeed shown that MAP below 65 mmHg, especially for extended periods, increases the risk of PMI.
* However, recent research is starting to challenge this perspective. Some studies have found that even maintaining a relatively higher blood pressure during surgery (e.g., MAP above 75 mmHg) didn't significantly reduce the incidence of PMI. This suggests that simply looking at a fixed blood pressure number might not tell the whole story.

Our preliminary research uncovered an intriguing finding: even if a patient's absolute blood pressure value during surgery seemed acceptable (e.g., above 60 mmHg), their risk of postoperative myocardial injury significantly increased if that pressure had dropped by more than 40% from their individual "normal" pre-operative blood pressure. Based on this discovery, our study proposes a novel hypothesis: the percentage drop in MAP from an individual's baseline might be more strongly correlated with postoperative myocardial injury and a better predictor of risk than the absolute MAP value.

The investigators will be reviewing patient data from non-cardiac surgeries performed at China-Japan Friendship Hospital between 2020 and 2025. The investigators will meticulously analyze these patients' intraoperative blood pressure changes (considering both absolute values and the percentage change from their pre-operative baseline) and compare these findings with whether they developed myocardial injury after surgery.

Our study's goal is to determine which definition of low blood pressure (absolute value or percentage drop from baseline) is more closely related to postoperative myocardial injury.

The investigators will collect detailed patient information, including demographics, past medical history, pre- and post-operative test results, intraoperative vital signs (blood pressure, heart rate, oxygen saturation, etc., recorded every 15 seconds), and intraoperative medications. All data will undergo rigorous statistical analysis to ensure the scientific validity and reliability of our findings.

The results of this study will help us more accurately identify patients at high risk for postoperative myocardial injury. If our hypothesis is confirmed, it means that during surgery, doctors, in addition to monitoring absolute blood pressure values, will pay closer attention to the degree of blood pressure drop relative to a patient's own normal baseline. This will help to:

* Improve understanding of individual patient differences: Recognizing that what's "normal" for one patient might be too low for another.
* Enable more precise adjustments in anesthesia and surgical management: Allowing for timely interventions to maintain optimal heart muscle perfusion, thereby reducing the incidence of postoperative myocardial injury.
* Ultimately, enhance patient safety during surgery and improve their recovery and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent elective non-cardiac, non-emergency surgery with general anesthesia at China-Japan Friendship Hospital between 2020 and 2025.
2. Surgical duration greater than 1 hour.
3. Received at least one cardiac injury marker test (e.g., troponin) within 7 days post-surgery.
4. Patients with American Society of Anesthesiologists (ASA) physical status classification of I-III.

Exclusion Criteria:

1. Patients younger than 12 years old.
2. Patients undergoing organ transplant surgery.
3. Patients with more than 10 consecutive minutes of invalid or missing intraoperative vital signs data.
4. Patients with critical missing data that cannot be reasonably imputed (general data completeness issues).

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study retrospectively includes adult patients (aged 12 years and older) who underwent elective, non-cardiac, non-emergency surgery under general anesthesia at China-Japan Friendship Hospital between January 2020 and December 2025. All included patients had a surgical duration exceeding 1 hour and an American Society of Anesthesiologists (ASA) physical status classification of I to III. A key criterion for inclusion was the availability of at least one cardiac injury marker test within 7 days post-surgery for outcome assessment. Patients undergoing organ transplant surgery or those with significant periods of missing or invalid intraoperative vital signs data (more than 10 consecutive minutes) will be excluded. The study cohort is expected to consist of approximately 8,000 patients, from whom detailed intraoperative hemodynamic data, patient demographics, comorbidities, surgical characteristics, and postoperative outcomes will be extracted for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
occurrence of postoperative myocardial injury | Within 7 days following non-cardiac surgery
  PMI is defined as an elevation of cardiac troponin (e.g., high-sensitivity troponin I or T) levels above the 99th percentile upper reference limit (URL) of the local institutional laboratory within 7 days following non-cardiac surgery. This outcome will be assessed based on routine postoperative cardiac biomarker measurements performed as part of standard clinical care. PMI serves as a critical indicator for evaluating cardiac damage post-surgery and is closely associated with adverse patient outcomes and prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- China-japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT07094321/Prot_SAP_000.pdf